CLINICAL TRIAL: NCT01041209
Title: Efficacy of BPS (Bacterial Pneumonia Score) Guided Antibiotic Use in Children With Community Acquired Pneumonia on Reducing Antibiotic Use as Compared to Standard Care Practice (Current Guidelines for CAP)
Brief Title: Bacterial Pneumonia Score (BPS) Guided Antibiotic Use in Children With Community Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HGNPE-186
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2013-06

CONDITIONS: Pneumonia
Keywords: Pneumonia; Children
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BPS (Experimental): BPS guidance
  Interventions: Behavioral: Strategy based on BPS guided antibiotic use
- Guideline (Active Comparator): Enforced guidelines
  Interventions: Behavioral: Enforced Guidelines

INTERVENTIONS:
Behavioral: Strategy based on BPS guided antibiotic use — In this study a strategy based on BPS guided antibiotic use in children with community acquired pneumonia implementation will be compared with enforced guideline.
  Arms: BPS
Behavioral: Enforced Guidelines — In this study a strategy based on BPS guided antibiotic use in children with community acquired pneumonia implementation will be compared with enforced guideline.
  Arms: Guideline

SUMMARY:
The aim of this study is to test if BPS (Bacterial Pneumonia Score) guided antibiotic use in children with non severe community acquired pneumonia (CAP) will reduce antibiotic use as compared to standard care practice (current guidelines for CAP).

DETAILED DESCRIPTION:
Background: Pneumonia is a leading cause of mortality in children. Despite more than 50% of pneumonias are due to viruses, because it is difficult to rule out bacterial etiology, initial management of pneumonia in children usually includes antibiotics, often unnecessary. In 2006 was designed and validated a clinical prediction rule (BPS: Bacterial Pneumonia Score) which accurately identifies hospitalized children's risk of bacterial pneumonia. However, BPS efficacy on guiding therapeutic decision in children with community acquired pneumonia (CAP) has not been yet assessed.

Aim: The aim of this study is to test if BPS guided antibiotic use in children with non severe community acquired pneumonia will reduce antibiotic use as compared to standard care practice (current guidelines for CAP) Design: This is a randomized, controlled, blinded trial, to assess antibiotics use regarding two methods for initial management of children aged 3-60 months with non severe community acquired pneumonia. Children will be randomly allocate to be managed according to BPS or currently enforced guidelines. Use of antibiotics (%) and clinical outcome of both groups will be compared.

Setting: Tertiary children hospital in Buenos Aires, Argentina. Patients: Consecutive children aged 3-60 months assisted for non severe community acquired pneumonia as outpatients. Patients with wheezing, severe pneumonia, pulmonary or cardiovascular chronic disease, or antibiotic use or hospitalization in the previous two weeks will be excluded.

Endpoints:

Primary: Use of antibiotics in each group (proportion) Secondary: Treatment failure (proportion) in each group Endpoints will be assessed at baseline and after 1, 2, 5, 7 and 10 days by a blinded investigator.

Intervention: Patients with CAP will be randomized (1:1) to BPS versus enforced guidelines. In the BPS group antibiotics will be indicated in patients with a BPS ≥ 4 points, while in the control group antibiotics will be indicated according to current guidelines.

Variables and measurement: Antibiotic use will be defined as initial use of any antibiotic, immediately after diagnosis. Treatment failure will be defined as persistence of fever after 2 days, or tachypnea or diminishing in respiratory rate less than 5 bpm. after 2 days, or signs of severe pneumonia or requiring or changing antibiotics at any time.

Study hypothesis: BPS antibiotic use guidance will reduce at least 20% antibiotic use, as compared to standard care practice.

Analyses: These will be done based on an intention-to-treat and a per-protocol principle. With an assumed 20% less use of antibiotics in the intervention group, a maximum of 5% losses to follow-up, a confidence of 5% and power of 90%, the total sample size is 60. This will allow detecting a difference in clinical outcome of 28%. Proportion will be compared by Chi square test.

Interim monitoring: Regular review of serious adverse events, quality and integrity of the study by an independent data safety and monitoring board. Safety interim analysis after 50% of the patients recruited.

Significance: Due to the high prevalence of CAP in children, this study will offer the potential for a substantial reduction in health costs and antibiotics resistance.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-60 months assisted as outpatients for non severe community acquired pneumonia.

Exclusion Criteria:

* Wheezing
* Severe pneumonia
* Pulmonary or cardiovascular chronic disease
* Antibiotic use in the previous two weeks
* Hospitalization for any reason in the previous two weeks

Ages: 3 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando A Torres, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de Niños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Moreno L, Krishnan JA, Duran P, Ferrero F. Development and validation of a clinical prediction rule to distinguish bacterial from viral pneumonia in children. Pediatr Pulmonol. 2006 Apr;41(4):331-7. doi: 10.1002/ppul.20364. PMID 16493666
- [Background] Ferrero F, Torres F, Noguerol E, Gonzalez N, Lonegro L, Chiolo MJ, Ossorio MF, Benguigui Y. [Evaluation of two standardized methods for chest radiographs interpretation in children with pneumonia]. Arch Argent Pediatr. 2008 Dec;106(6):510-4. doi: 10.1590/S0325-00752008000600007. Spanish. PMID 19107303
- [Result] Torres FA, Pasarelli I, Cutri A, Ossorio MF, Ferrero F. Impact assessment of a decision rule for using antibiotics in pneumonia: a randomized trial. Pediatr Pulmonol. 2014 Jul;49(7):701-6. doi: 10.1002/ppul.22849. Epub 2013 Aug 23. PMID 24039234

RESULTS

PARTICIPANT FLOW:
Groups:
- Bacterial Pneumonia Score (BPS): Use of antibiotics according to Bacterial Pneumonia Score (BPS) guidance (antibiotic use when BPS > or = 4 points)
- Guideline: Use of antibiotics according to local enforced guidelines
Period: Overall Study
Arm/Group | Bacterial Pneumonia Score (BPS) | Guideline
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bacterial Pneumonia Score (BPS): Bacterial Pneumonia Score (BPS) guidance
- Total: Total of all reporting groups
Arm/Group | Bacterial Pneumonia Score (BPS) | Guideline | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 120
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (13.2) | 26.1 (13.2) | 24.2 (14.1)
Gender [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 27 | 30 | 57
Region of Enrollment [Number; unit: participants]
  Argentina | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Use of Antibiotics in Each Group
Description: The proportion of patients receiving antibiotics was compared between both groups (BPS vs Guidelines).
Time Frame: At baseline
Measure: Number; unit: participants
Groups:
- Bacterial Pneumonia Score (BPS): Indication of antibiotics according to Bacterial Pneumonia Score (BPS) guidance. Antibiotics were indicated with BPS >= 4 points
- Guideline: Indication of antibiotics according to local (Hospital) guidelines
Arm/Group | Bacterial Pneumonia Score (BPS) | Guideline
Number analyzed (Participants) | 60 | 60
participants | 28 | 52

2. Secondary Outcome: Treatment Failure in Each Group
Description: Treatment failure was defined as: Persistence of fever after 2 days, or tachypnea or diminishing in respiratory rate less than 5 bpm after 2 days, or signs of severe pneumonia or requiring or changing antibiotics at any time.
  Proportion of patients with treatment failure was compared between both groups (BPS vs Guideline).
Time Frame: 1, 2, 5, 7 and 10 days from baseline
Measure: Number; unit: participants
Groups:
- Guideline: Indication of antibiotics according to local (Hospital)guidelines.
Arm/Group | Bacterial Pneumonia Score (BPS) | Guideline
Number analyzed (Participants) | 60 | 60
participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Bacterial Pneumonia Score (BPS) | Guideline
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes